CLINICAL TRIAL: NCT03309995
Title: The Effect of Zinc Acetate Lozenges on the Rate of Recovery From the Common Cold: a Randomized Trial
Brief Title: The Effect of Zinc Acetate Lozenges on the Rate of Recovery From the Common Cold
Acronym: HelZinki
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Helsinki (Other)
Collaborators: The University Pharmacy, Helsinki (Unknown)
Responsible Party: Principal Investigator, Harri Hemilä, MD, PhD, Senior researcher, docent, University of Helsinki
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: HelZinki Study
Record Dates: First submitted 2017-10-10; First posted 2017-10-16 (Actual); Last update posted 2020-02-05 (Actual); Status verified 2020-01

CONDITIONS: Common Cold; Respiratory Tract Infections
Keywords: Cough; Laryngitis; Pharyngitis; Rhinitis; Zinc Acetate; Zinc Lozenge
MeSH Terms: conditions — Common Cold; Respiratory Tract Infections; Cough; Laryngitis; Pharyngitis; Rhinitis | interventions — Tobacco Use Cessation Devices

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Zinc lozenges (Experimental): Each lozenge contains 13 mg elemental zinc as zinc acetate. The instruction for common cold patients is to dissolve slowly 6 lozenges per day in their mouth, which totals to 78 mg/day of elemental zinc, at most for 5 days, as early as possible from the start of the cold symptoms.
  Interventions: Device: Lozenges
- Placebo lozenges (Placebo Comparator): The placebo lozenges contain sucrose octaacetate, and they are similar with the zinc lozenges in visual appearance and in taste.
  Interventions: Device: Placebo lozenges

INTERVENTIONS:
Device: Lozenges — The participants will be instructed to take 6 lozenges daily over the time awake, evenly distributed, allowing the lozenge to dissolve in the mouth as slowly as possible.
  Arms: Zinc lozenges
Device: Placebo lozenges — Placebo lozenges
  Arms: Placebo lozenges

SUMMARY:
A randomized parallel-group two arm superiority trial with an allocation ratio 1:1, both participants and investigators blinded.

The zinc lozenge that will be used in the study is a commercial product available from the University Pharmacy, Helsinki, Finland. The product is classified as a "medical device" and it is not regulated according to the jurisdiction for medicines.

Each lozenge contains 13 mg elemental zinc as zinc acetate. The instruction in the commercial package for common cold patients is to dissolve slowly 6 lozenges per day in their mouth, which totals to 78 mg/day of elemental zinc, at most for 5 days. The same instruction will be used in this trial.

The University Pharmacy prepared 200 placebo lozenge packages so that the placebo lozenges contain sucrose octaacetate, and they are similar with the zinc lozenges in visual appearance and in taste. 200 packages of zinc lozenges will be used as the active intervention. The packages will contain 30 lozenges (6 lozenges/day × 5 days).

The packages of lozenges will be distributed to the enrolled participants in November 2017. The participants will be instructed to keep the package readily available so that, when they catch the common cold, they will find the package and they can start to take the lozenges according to the instructions.

The participants will be instructed to start taking zinc lozenges as soon as they start to suffer from the first symptoms of the common cold. The participants will be instructed to take 6 lozenges daily over the time awake, evenly distributed, allowing the lozenge to dissolve in the mouth as slowly as possible. The duration of intervention is for the maximum of 5 days. If the symptoms disappear before 5 days, the participant may stop the usage of the lozenges.

There will be no limitations for other treatments that participants wish to use for treating their colds.

Participants will be requested to respond to a web-based symptom questionnaire daily from the first day of the treatment to the recovery from the common cold, or to a maximum of 2 weeks.

ELIGIBILITY:
Inclusion Criteria:

* ≥18 years, recollecting that they usually have had ≥1 colds per winter.

Exclusion Criteria:

* pregnancy or lactation; chronic runny nose or chronic cough.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 87 (Actual)
Dates: Start 2017-12-01 (Actual); Primary Completion 2018-04-24 (Actual); Study Completion 2018-09-24 (Actual)

PRIMARY OUTCOMES:
The duration of the common cold (time to recovery) | 2 weeks after the start of the intervention
  Data of 12 common cold symptoms will be recorded by patients to web-based system, with scale 0: Absent, 1: Mild, 2: Moderately severe, 3: Very severe symptom. The symptom score is calculated as a sum over all the symptoms which means that the maximum of the symptom score scale is 3×12 = 36 points. Recovery from the cold is defined as the day when the symptom score is 0 or 1.

SECONDARY OUTCOMES:
Objective fever | 2 weeks after the start of the intervention
  Measured fever (≥37.5°C any time during the day) (Yes / No)
Sickness absence | About 1 month after the start of the intervention
  Data will be collected of the absence from work after the start of intervention
Usage of antibiotics and/or asthma medication | About 1 month after the start of the intervention
  Data will be collected of the usage of antibiotics and/or asthma medication after the start of intervention
Complications such as sinusitis, bronchitis, otitis. | About 1 month after the start of the intervention
  Data will be collected of the occurrence of sinusitis, bronchitis, otitis after the start of intervention

CONTACTS AND LOCATIONS:
Overall Officials: Harri Hemilä, MD, PhD, Principal Investigator — University of Helsinki
Locations (1):
- City of Helsinki, Helsinki, Finland

IPD SHARING:
Plan to Share IPD: Yes
IPD reported with the trial report (2020)
Time Frame: Upon the publication of trial report indefinitely
Access Criteria: IPD reported with the trial report (2020) is freely available

REFERENCES:
- [Result] Hemila H, Haukka J, Alho M, Vahtera J, Kivimaki M. Zinc acetate lozenges for the treatment of the common cold: a randomised controlled trial. BMJ Open. 2020 Jan 23;10(1):e031662. doi: 10.1136/bmjopen-2019-031662. PMID 31980506
- See also: Report of the trial — http://dx.doi.org/10.1136/bmjopen-2019-031662